CLINICAL TRIAL: NCT04578691
Title: A Two-arm, Single Center, Randomised Study to Evaluate the Safety and Clinical Outcome of Using Navigation System in Pedicle Screw Placement in Spine Surgery
Brief Title: Study to Evaluate the Safety and Clinical Outcome of Using Navigation System in Pedicle Screw Placement in Spine Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Taipei Veterans General Hospital, Taiwan (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2020-03-004C
Record Dates: First submitted 2020-08-20; First posted 2020-10-08 (Actual); Last update posted 2022-11-10 (Actual); Status verified 2022-11

CONDITIONS: Spinal Tumor; Traumatic Injury of Spine; Degenerative Spine Disease
Keywords: Pedicle screw placement surgery; 10th thoracic vertebra to 1st sacrum
MeSH Terms: conditions — Spinal Cord Neoplasms; Spinal Injuries

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- "Anatase" Spine Surgery Navigation System (Experimental): Using "Anatase" Spine Surgery Navigation System in pedicle screw placement in spine surgery
  Interventions: Device: "Anatase" Spine Surgery Navigation System
- Medtronic Stealthstation S7 Treatment Guidance System (Active Comparator): Using Medtronic Stealthstation S7 Treatment Guidance System in pedicle screw placement in spine surgery
  Interventions: Device: Medtronic Stealthstation S7 Treatment Guidance System

INTERVENTIONS:
Device: "Anatase" Spine Surgery Navigation System — using navigation system in pedicle screw placement in spine surgery
  Arms: "Anatase" Spine Surgery Navigation System
Device: Medtronic Stealthstation S7 Treatment Guidance System — using navigation system in pedicle screw placement in spine surgery
  Arms: Medtronic Stealthstation S7 Treatment Guidance System

SUMMARY:
The research project is testing whether in screw insertion of spine surgery using "Anatase" Spine Surgery Navigation System is at least as safe and accurate as using O-arm assisted spine surgery- Medtronic Stealthstation S7 Treatment Guidance System.

DETAILED DESCRIPTION:
Pedicle screw insertion is performed to treat the patients with spine conditions, including degenerative, traumatogenic, and neoplastic lesions. Accurate insertion of pedicle screw is a crucial step which directly affects the surgical outcomes. In order to place the screws safely and accurately, various conventional techniques have been used, focusing on marking anatomical locations, entry points and insertion angles. Since the early 1990, the methods using computer systems that allow real-time image processing have been explored in order to improve the accuracy of pedicle screw placement.

The Medtronic StealthStation® S7® System is a hardware platform that enables real-time surgical navigation using radiological patient images. The application software reformats patient-specific CT or MR images acquired before surgery, or fluoroscopic images acquired during surgery, and displays them on-screen from a variety of perspectives. The "Anatase" Spine Surgery Navigation System is indicated for precisely positioning of surgical instruments and/or implants during general spinal surgery, such as pedicle screw placement.

This study will be a two-arms, single center, evaluator blind, controlled, parallel, randomised study in patients with pedicle screw placement in spine surgery. This trial will include patients need to undergo pedicle screw placement surgery with indication of spinal tumor, traumatic injury or degenerative spine disease (Pedicle screws placed from 10th thoracic vertebra to first sacrum), who are ≥20 years and ≤80 years of age with Body Mass Index (BMI) < 40 kg/m2 and Spine T-Score ≥ -2.5.

ELIGIBILITY:
Inclusion Criteria:

1. Patients who need to undergo pedicle screw placement surgery with indication of spinal tumor, traumatic injury or degenerative spine disease.
2. Pedicle screws placed from 10th thoracic vertebra to first sacrum.
3. Age ≥20 years and ≤80 years.
4. Body Mass Index (BMI) < 40 kg/m2.
5. Spine T-Score by Dual Energy X-ray Absorptiometry ≥ -2.5, 60 days prior to surgery.
6. The subject is willing and able to comply with the procedure and requirements of this trial.
7. The participant is able to understand and provide informed consent, and has signed their written informed consent in accordance with IRB requirements.

Exclusion Criteria:

1. Pregnant women.
2. Hereditary or acquired haemorrhagic diathesis or coagulation factor deficiency.
3. Be on uncontrolled Diabetes mellitus.
4. Any history of stroke within the previous 6 months.
5. Any history or current evidence suggestive of Coronary Artery Disease or Cerebral Vascular Accident within the previous 6 months, including clinical, EKG, laboratory, or imaging findings.
6. Any terminal illness such that the patient would not be expected to survive more than 6 months.
7. Creutzfeldt-Jakob disease.
8. Known allergy to stainless steel (device material).
9. Have a systematic or local infection, which may increase study risk.
10. Immunocompromised such as but not limited to Acquired Immunodeficiency Syndrome (AIDS), HIV infection, Severe Combined Immunodeficiency Syndrome, Thymic Hypoplasia.
11. Immunologically suppressed, or has received systemic steroids, excluding nasal steroids, at any dose daily for > 1 month within last 12 months.
12. Any condition that, in the judgment of the investigator, could impose hazards to the patient if study therapy is initiated or affect the participation of the patient in the study.
13. Former spinal surgery may interfere with the present trial.
14. Participation in any investigational study in the last 30 days or current enrolment in any trial. Non- interventional Studies are not considered exclusion.
15. Any condition that increases anesthesia risk.

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 55 (Actual)
Dates: Start 2020-06-29 (Actual); Primary Completion 2022-06-03 (Actual); Study Completion 2022-08-31 (Actual)

PRIMARY OUTCOMES:
Rate of screw outside the vertebral body | not later than discharge, up to 14 days
  Rate of screw outside the vertebral body as measure by post CT image which perform not later than discharge.

SECONDARY OUTCOMES:
Difference between the actual and virtual (navigation image) of screw's sharp point position | not later than discharge, up to 14 days
  Blind Assessor will measure the distance (mm) between the actual (post-CT) and virtual (baseline CT) of screw's sharp point position.
Difference between the actual and virtual (navigation image) angle of screws | not later than discharge, up to 14 days
  Blind Assessor will measure the difference of angle (°) between the actual (post-CT) and virtual (baseline CT)screws.
Blood loss during surgery (mL) | operation 1 day
  record the blood loss during surgery (mL)
Total intraoperative radiation exposure for the operator and patient | 1 day, the TLD badges will be detected
  Record the total intraoperative radiation exposure of operator and patient wearing TLD badges
Mean time required for preparation of screw placement (min) | operation 1 day
  Record the mean time required for preparation of screw placement (min)
Time to accomplish each screw insertion (min) | operation 1 day
  Record the time to accomplish each screw insertion (min)
Ratio of revision surgery within 3 months after main surgery | after 3 months of surgery
  Record ration of revision surgery within 3 months after main surgery
Length of postoperative hospital stay | Discharge day, up to 14 days
  Record length of postoperative hospital stay
Adverse event (AE) and serious AE (SAE) incidence rates during the trial | 90 days
  Record Adverse event (AE) and serious AE (SAE) during the trial

CONTACTS AND LOCATIONS:
Overall Officials: Tsung-Hsi Tu, Principal Investigator — Taipei Veterans General Hospital, Taiwan
Locations (1):
- Taipei Veterans General Hospital, Taipei, Taiwan

IPD SHARING:
Plan to Share IPD: No